CLINICAL TRIAL: NCT01477086
Title: Prevalence and Pathophysiology of Sarcopenia in the Elderly Patient With Hip Fracture. Prospective, Observational Study on Consecutive Series
Brief Title: Prevalence and Pathophysiology of Sarcopenia in the Elderly Patient With Hip Fracture
Acronym: PREFISSARC
Status: Completed | Type: Observational
Sponsor: Hospital Viamed Valvanera, Spain (Other)
Collaborators: University of Navarra (Other)
Responsible Party: Sponsor
Other Study IDs: Viamed-Sarco-HF
Record Dates: First submitted 2011-10-19; First posted 2011-11-22 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Sarcopenia; Hip Fracture; Frailty
Keywords: Sarcopenia; Hip fracture; Frailty
MeSH Terms: conditions — Sarcopenia; Hip Fractures; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hip fracture: We included patients with traumatic hip fracture, with surgery and who are admitted for rehabilitation

SUMMARY:
Sarcopenia is the loss of muscle mass and function that accompanies aging. The term sarcopenia comes from the Greek "sarx" (flesh) and "penia" (loss).

Sarcopenia is a topic of great interest to geriatricians, and from 2010 discussing the possibility of considering it as a geriatric syndrome.

Diagnostic criteria are reduced muscle mass, reduced strength and impaired physical performance. The presence of muscle mass reduction set presarcopenia diagnosis, when combined with one of the other two are talking about sarcopenia and when are the three is defined as severe sarcopenia.

The hypothesis of our study is that sarcopenia is highly prevalent in older people with hip fracture. The increase in inflammatory indices of older people, along with bed rest, represent factors that accelerate the development of sarcopenia. These factors together could be the base of the high percentage of patients who do not recover the degree of autonomy before the fracture.

DETAILED DESCRIPTION:
The incidence of hip fracture in Spain is estimated at 551 cases per 100,000 population aged 65 years, with an average cost of treatment for a broken € 9,996.00 and more days of hospitalization than heart attacks. In-hospital mortality is 5.3%. Data from a multicenter study in 77 hospitals of the Spanish territory in 2003 coincide with those of studies conducted in other European countries regarding the incidence, the highest percentage in women and increased exponentially with age.

The fracture of the proximal femur (hip) is a substantial cause of morbidity and mortality in the elderly. Mortality at one year after hip fracture varies between 12 and 37%, with an incidence of 11% during the first months.

25% of elderly patients with hip fracture requires institutionalization, at least temporarily, and only 40% fully recover their functional status before the fracture.

Hip fracture is a major public health problem. It happens more often in the elderly, the average age of patients admitted is 81.4 ± 8.1 years and its incidence has increased significantly in recent years. It causes a high degree of disability, mortality and frequent large economic costs. 50% of patients independent before a hip fracture are unable to recover fully the functionality, face and often the inability to institutionalization.

Only 30-35% of elderly hip fractures regain their previous degree of independence in basic activities of daily living, and only 20-25% do so for instrumental activities.

The investigators hope to find a high prevalence of sarcopenia in patients admitted with hip fracture, and patients with more severe sarcopenia are those having lower functional levels at admission and discharge phenomenon recover. The investigators hope to find a relationship between elevated inflammatory indices and severity of sarcopenia. The investigators hope that the presence of sarcopenia, and its severity, correlates positively with the occurrence of complications during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 65 years;
* Diagnosis of traumatic fracture of hip;
* To sign informed consent (patient or legal guardian, if cognitive impairment).

Exclusion Criteria:

- Excluding patients will not sign the informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Will be included in the study, prospectively, patients with hip fracture admitted to the Geriatric Rehabilitation Unit, Spain.
Sampling Method: Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2012-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Sarcopenia prevalence | Within the first 72 hours of admission.
  To study the prevalence of sarcopenia in patients with hip fracture, those are hospitalized for rehabilitation. For the diagnosis of sarcopenia will use the criteria of the EWGSOP (1). Will be used bioelectrical impedance (BIA).For the BIA, we use the cut-off proposed by Jansen (2).

SECONDARY OUTCOMES:
Relationship inflammatory indices and sarcopenia. | A admission and at discharge, after 30 days.
  To demonstrate whether patients with sarcopenia are those with higher levels of inflammatory markers. By measurements of IL-1, IL-6, TNF-alpha and acute phase proteins at admission and at discharge, expected average of 30 days.
Prevalence of falls. | During the six months prior to admission.
  Will record the number of falls, with and without consequences, in the six months prior to admission.
Acute mortality. | During admission
  Relation between mortality from any cause and sarcopenia. Correcting the statistical analysis for confounding factors.
Relationship sarcopenia and frailty. | At admission and after 30 days.
  Relating the results of bioelectrical impedance and fragility. For the diagnosis of frailty we will refer to the original criteria proposed by L. Fried (3). participants will be followed for the duration of hospital stay, an expected average of 4 weeks
Relationship sarcopenia and Barthel index. | At admission and after 30 days .
  Demonstrate that patients with sarcopenia are those with more functional limitations after rehabilitation. By contrast to the Barthel index at admission and at discharge, expected average of 30 days of rehabilitation, and the difference between the Barthel Index before fracture and at discharge. The assessment of functional limitation will be performed with the validated Spanish version of the SF-LLDFI (7).

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Malafarina, MD MSc, Principal Investigator — Clinica Los Manzanos, Lardero, Spain
Locations (1):
- Hospital Viamed Valvanera, Logroño, La Rioja, Spain

REFERENCES:
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Janssen I. Influence of sarcopenia on the development of physical disability: the Cardiovascular Health Study. J Am Geriatr Soc. 2006 Jan;54(1):56-62. doi: 10.1111/j.1532-5415.2005.00540.x. PMID 16420198
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Perez Durillo FT, Ruiz Lopez MD, Bouzas PR, Martin-Lagos A. [Nutritional status in elderly patients with a hip fracture]. Nutr Hosp. 2010 Jul-Aug;25(4):676-81. Spanish. PMID 20694307
- [Background] Herrera A, Martinez AA, Ferrandez L, Gil E, Moreno A. Epidemiology of osteoporotic hip fractures in Spain. Int Orthop. 2006 Feb;30(1):11-4. doi: 10.1007/s00264-005-0026-2. Epub 2005 Nov 18. PMID 16328387
- [Background] Roberts HC, Denison HJ, Martin HJ, Patel HP, Syddall H, Cooper C, Sayer AA. A review of the measurement of grip strength in clinical and epidemiological studies: towards a standardised approach. Age Ageing. 2011 Jul;40(4):423-9. doi: 10.1093/ageing/afr051. Epub 2011 May 30. PMID 21624928
- [Background] Abizanda P, Lopez-Jimenez M, Lopez-Torres J, Atienzar-Nunez P, Naranjo JM, McAuley E. Validation of the Spanish version of the Short-Form Late-Life Function and Disability Instrument. J Am Geriatr Soc. 2011 May;59(5):893-9. doi: 10.1111/j.1532-5415.2011.03392.x. PMID 21568958
- [Background] Malafarina V, Uriz-Otano F, Iniesta R, Gil-Guerrero L. Sarcopenia in the elderly: diagnosis, physiopathology and treatment. Maturitas. 2012 Feb;71(2):109-14. doi: 10.1016/j.maturitas.2011.11.012. Epub 2011 Dec 6. PMID 22153348
- [Background] Malafarina V, Uriz-Otano F, Iniesta R, Gil-Guerrero L. Effectiveness of nutritional supplementation on muscle mass in treatment of sarcopenia in old age: a systematic review. J Am Med Dir Assoc. 2013 Jan;14(1):10-7. doi: 10.1016/j.jamda.2012.08.001. Epub 2012 Sep 13. PMID 22980996